CLINICAL TRIAL: NCT07351123
Title: Assessment of Treatment Variability for Pelvic Ring Fragility Fractures
Acronym: Pelvis ATV
Status: Not yet recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Mark Gage, Associate Professor, University of Maryland, Baltimore
Other Study IDs: 1R01AR086467-01 (NIH); 1R01AR086467-01 (NIH)
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Fractures; Fragility Fractures of the Pelvis (FFP)
Keywords: Pelvic fracture; Fragility fracture of the pelvis; Pelvic ring injury
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients aged 60 years and older with a low energy mechanism closed pelvic ring fracture with an anterior and posterior injury observable on x-ray or CT scan
  Interventions: Procedure: Surgical stabilization of pelvic fracture; Other: Closed treatment of pelvic fracture

INTERVENTIONS:
Procedure: Surgical stabilization of pelvic fracture — Surgical stabilization of pelvic fracture through placement of orthopaedic hardware.
Other: Closed treatment of pelvic fracture — Pelvic fracture that is treated without surgery and assessed over time through interval radiographs until fracture is healed.

SUMMARY:
Fragility fractures of the pelvic ring are a common injury associated with poor patient outcomes and high healthcare costs. Management of these injuries is evolving with increasing frequency of operative stabilization of the pelvic ring, despite a lack of evidence supporting operative versus nonoperative treatment. This multicenter prospective cohort study will evaluate 120 patients to determine the feasibility of a randomized controlled trial comparing operative and nonoperative treatment, by evaluating patient willingness to enroll in a trial, surgeon willingness to randomize their patients' treatment, and the completeness of data collection.

DETAILED DESCRIPTION:
Fragility fractures of the pelvic ring are a common injury that is increasing in incidence with an aging population. These injuries are associated with high healthcare costs and poor patient outcomes, including decline in ambulatory function, decreased independence, and a one-year mortality of 11-27%. Historically, older adults with fragility fractures of the pelvis received nonoperative treatment with supportive care because operative management was deemed too invasive for this patient population. However, the development of percutaneous and less invasive surgical techniques has led to an increased frequency of operative stabilization of pelvis fractures in older adults. It is unclear if the increasing use of surgical fixation is improving outcomes for patients with pelvic fragility fractures. There are significant limitations with the current body of evidence that precludes its ability to guide clinical practice. Randomized controlled trials testing the efficacy of operative management are urgently needed to determine when surgical fixation is warranted.

Two pilot randomized controlled trials have been performed on this patient population, and both have not progressed to a definitive study citing a lack of recruitment feasibility. This is due to both the lack of agreement amongst surgeons for which patients should receive randomized treatment, as well as a lack of patient willingness to enroll in a trial. Furthermore, loss to follow up is a concern in both the orthopaedic trauma population and in older adult study patients. This prospective cohort study will evaluate 120 patients from six hospitals to determine the feasibility of a randomized controlled trial (RCT) comparing operative versus nonoperative management of fragility fractures of the pelvic ring. This will be accomplished by three aims evaluating patient willingness to enroll in a trial, surgeon willingness to randomize their patients' treatment, and the completeness of data collection.

ELIGIBILITY:
The inclusion criteria are:

1. Patient 60 years of age or older.
2. Low energy injury mechanism.
3. LC1 pelvis fracture (AO/OTA 61B1.1,61B2.1, or 61B3.2) confirmed with antero-posterior, inlet, and outlet pelvis radiographs, computed tomography, or magnetic resonance imaging.
4. Fracture displacement of <10 mm of the posterior pelvic ring on computed tomography of the pelvis.
5. Injury occurred within 21 days of screening.

The exclusion criteria are:

1. Patient did not ambulate prior to injury.
2. Severely frail patients (Clinical Frailty Scale ≥7).
3. Patient has another condition, injury, or fracture that prevents post-operative weightbearing on any extremity.
4. Retained implants around the pelvis that precludes or limits either study treatment.
5. Infection around the hip (soft tissue or bone).
6. Pathologic fracture with a lytic lesion in the pelvis or sacrum that precludes internal fixation.
7. Patient is too ill, in the judgement of the attending surgeon, for internal fixation.
8. Patient is too ill, in the judgement of the attending surgeon, for nonoperative care.
9. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
10. Expected injury survival of less than 12 months.
11. Terminal illness with expected survival of less than 12 months.
12. Currently enrolled in a study that does not permit co-enrollment.
13. Prior enrollment in the study.
14. Unable to obtain informed consent due to language barriers.
15. Unable to obtain informed consent because a legally authorized representative (LAR) was unavailable.
16. Did not provide informed consent (declined participation).
17. Patient or LAR not approached to participate in the trial (missed patient).
18. Other reason to exclude the patient, as approved by the Principal Investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 60 years of age with a closed pelvic ring fracture with an anterior and posterior injury observable on x-ray or CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Willingness to Enroll in a Trial | 4 months
  Willingness to enroll in a trial will be assessed as a binary variable with the central three choices representing that the participant is willing to have their treatment randomized.
Surgeon Willingness to Randomize Patient Treatment | 4 months
  Surgeon willingness to enroll the patient in the trial will be assessed as a binary variable with the central three choices representing that the surgeon would have been willing to have their treatment decision randomized.
Completeness of Patient Centered Outcomes Collected | 4 months
  The outcome measure completion will be assessed as a binary variable classified as either complete documentation or missing documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gage, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: Yes
The Final Research Data set of validated de-identified data will include discrete data elements supporting the primary and secondary endpoints. Demographic, injury, clinical results data will be acquired from pelvis fracture subjects. All data will be de-identified prior to receipt by the National Trauma Research Repository (NTRR).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to the research community as soon as possible, but no later than one year after publication of the initial study manuscript. All data will be kept in the NTRR for at least five years after the initial study publication.
Access Criteria: All data and associated study materials will be submitted to the NTRR. The NTRR is built on the Biomedical Research Information Computing System (BRICS) platform developed by the Center for Information Technology at the National Institutes of Health (NIH). The NTRR platform and processes meet the NIH Grant Policy on Sharing of Unique Research Resources, including the Sharing of Biomedical Research Resources Principles and Guidelines for Recipients of the NIH Grants and Contracts.
  Data will be findable for the research community through the NTRR. The NTRR assigns a unique digital object identifier (DOI) for each data set submitted. This DOI, as a persistent unique identifier, can be used to reference the data set in manuscripts. Data stored in the NTRR meets FAIR principles (findable, accessible, interoperable, and re-usable).